CLINICAL TRIAL: NCT05020119
Title: A Phase I Study to Evaluate the Safety, Tolerability, and Antitumor Activity of Neoantigen-expanded Autologous Immune Cell Therapy for Solid Tumors
Brief Title: Neoantigen-expanded Autologous Immune Cell Therapy
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, HOU, MING-MO, Attending physician, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DC-CIK_TRIAL_PROPOSAL
Record Dates: First submitted 2021-07-30; First posted 2021-08-25 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Intervention Model Description: This study aims to investigate the safety profile and therapeutic potential of neoantigen-expanded autologous immune cell for treating solid tumors. The safety evaluation will be performed by a traditional 3+3 dose escalation scheme. The three cohorts will be established in the trial, and the dose level of each cohort will be enrolling 3~6 subjects.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low dose of neoantigen-based cell therapy (N=3+3) (Experimental): (1±20%) × 109cells/200 mL every 14 days for 10 doses
  Interventions: Drug: Neoantigen-expanded cell therapy.
- Medium dose of neoantigen-based cell therapy (N=3+3) (Experimental): (3±20%) × 109cells/200 mL every 14 days for 10 doses
  Interventions: Drug: Neoantigen-expanded cell therapy.
- High dose of neoantigen-based cell therapy (N=3+3) (Experimental): (9±20%) ×109cells/400 mL every 14 days for 10 doses
  Interventions: Drug: Neoantigen-expanded cell therapy.

INTERVENTIONS:
Drug: Neoantigen-expanded cell therapy. — Infusion of personalized neoantigen-expanded T (CIK) cells
  Other Names: Neoantigen-expanded autologous DC-CIK cells.

SUMMARY:
The investigators aim to investigate the patient's tumor neoantigen to generate "personalized cancer vaccine" and then to expand autologous dendritic cells-cytokine-induced killer cells (DC-CIK). The autologous DC-CIK will be cultured in vitro and re-infused into patients.

DETAILED DESCRIPTION:
Cancer is the leading cause of death in the world. However, the response of traditional treatments(such as chemotherapy, radiotherapy, or target therapy) is yet limited. In this clinical trial study, the investigators will investigate the patient's tumor neoantigen to generate "personalized cancer vaccine" and then to expand autologous dendritic cells-cytokine-induced killer cells (DC-CIK). The autologous DC-CIK will be cultured in vitro and re-infused into patients. The similar clinical trial design and immune cell preparation have been recently published in international journals. Though adverse reactions (AE) have been reported, and there was no cases with severe adverse events (SAE), suggesting the safety of autologous immune cell therapy against cancers. The main propose of this clinical trial is to improve the treatment for solid tumors. By conducting this clinical trial, the investigators aim to enroll patients with refractory advanced solid tumors, and develop "neoantigen-expanded autologous immune cell therapy". The investigators will utilize "neoantigens" to expand the patients' autologous peripheral blood mononuclear cells into DC-CIK. The enrolled patients will receive autologous DC-CIK of 10 doses within 4~5 months of treatment, and the safety, tolerability, and efficacy of this immune cell therapy will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. The patient has one of the following solid tumors, including colorectal cancer, gastric cancer, pancreatic cancer, esophageal cancer, liver cancer, gastrointestinal stromal tumor, biliary tract cancer, kidney cancer, bladder cancer, prostate cancer, Head and neck cancer, nasopharyngeal cancer, skin cancer, melanoma, malignant sarcoma, breast cancer, ovarian cancer, cervical cancer, endometrial cancer, lung cancer, and brain cancer.
2. The patient has at least one lesion that can be obtained by sectioning or cutting to identify somatic mutations from the tumor.
3. The patient diagnosed as advanced solid tumor is refractory to standard treatment; or intolerable to or unsuitable for standard treatment.When evaluating to participate in the trial, the patient must still have solid tumor.

   All patients are refractory to approved standard treatment.The definition of standard treatment for different cancers is listed below.
   1. Patient with colorectal cancer must have received surgery or at least two prior chemotherapies, including oxaliplatin and irinotecan; or at least one of the target therapies for colorectal cancer, including Cetuximab, Bevacizumab, Panitumumab, etc.
   2. Patient with gastric cancer and pancreatic cancer must have received radiotherapy, surgery, or received chemotherapies.
   3. Patient with esophageal cancer must have receivedthesecond-line systemic drug therapy (eg. chemotherapies or immunotherapies)
   4. Patient with liver cancer must havereceivedsurgery; radio-frequency ablation, or transcatheterial chemoembolization.
   5. Patient with biliary tract cancer must have refractory to the first-line treatment containing gemcitabine.
   6. Patient with gastrointestinal stromal tumors must have received the first-line target treatments.
   7. Patient with renal cancer must have received 2nd-line treatments (including chemotherapies or target therapies or combination with immunotherapies.
   8. Patient with bladder cancer must have received platinum-based chemotherapy or unable to receive chemotherapies and received immunotherapy.
   9. Patient with prostate cancer must have continued to disease progression or recur after receiving chemotherapies or the second-line hormone therapies.
   10. Patient with head and neck cancer and nasopharyngeal carcinoma must have received chemotherapies, including cetuximab or platinum.
   11. Patient with skin cancer and melanoma must have received at least one systemic treatment.

       If there is a genetic mutation for enrolled patients, the patient must be refractory to target therapies (related to mutation) or to the first-line chemotherapies.
   12. Patient with malignant sarcoma must have received first-line chemotherapies or target therapies.
   13. Patient with breast cancer who are unable to undergo surgery must have received anthracycline taxsnes and any third-line medication. If the patient with a positive ER gene, at least three third-line hormone therapies should be used. If patient with a positive HER2 gene, at least Hercrptin and Perjecta or T-DM1 should be used.
   14. Patient with ovarian cancer must have received platinum-containing chemotherapies to stop recurrence within 1-6 months; or have done more than the 2nd-line chemotherapies.
   15. Patient with cervical cancer must have received radiation therapy and chemotherapies.
   16. Patient with endometrial cancer must have received hormone therapy or radiotherapy.
   17. Patient with lung cancer must be refractory to the first-line standard treatment contained with platinum-based doublet chemotherapy in the patient without detected driver mutation or have failed to tyrosine kinase inhibitors and standard platinum-based doublet chemotherapy in those with drug related driver mutation.
   18. Patient with brain cancer must have received radiation therapy and chemotherapies; or patient's tumor still recurs within one to six months after chemotherapies, andcan not be completely resected; or patients have failed to target therapies.
4. The patient who is willing to receive cell therapy.
5. Age is greater than or equal to 20 years old.
6. Clinical performance status of ECOG 0 or 1.
7. Life expectancy exceeds six months
8. Patients can take foods and drugs orally.
9. Hematology:

   1. Absolute neutrophil count greater than 1000/mm3 without support of filgrastim
   2. Normal WBC (> 3000/mm3).
   3. Hemoglobin greater than 8.0 g/dl. Subjects may be transfused to reach this cut-off.
   4. Platelet count greater than 100,000/mm3
   5. Normal prothrombin time (less than or equal to 15.2 seconds)
10. The heart, lung and liver function of the patient must comply with:

    1. NYHA (the New York Heart Association) Functional Class I or II
    2. Serum ALT / AST is less than 150 U/L (patients with advanced hepatocellular carcinoma need to be less than 180 U/L)
    3. Serum creatinine less than or equal to 1.6 mg/dl.
    4. Total bilirubin less than or equal to 2 mg/dl, except in patients with Gilbert's Syndrome, who must have a total bilirubin less than or equal to 3 mg/dl.
    5. eGFR is greater than 60mL/min/1.73m2 (patients with advanced renal cell carcinoma need to be greater than 50 mL/min/1.73m2)
11. Patient with primary major surgery needs to have elapsed ≥ 4 weeks prior to the planned first study treatment day.
12. Patient who has ever received chemotherapy, radiotherapy or immunotherapy (anti-CTLA4 or anti-PD1/PDL1), or biologic therapy (anti-VEGF or anti-TKR) modalities need to washout ≥ 4 weeks prior to the baseline visit.
13. Stop receiving systemic immunosuppressive drugs within 7 days before starting the immune cell infusion
14. Willing to practice birth control during treatment
15. Able to understand and sign the Informed Consent form

Exclusion Criteria:

1. Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the treatment on the fetus or infant.
2. A systemic infections (e.g.: requiring anti-infective treatment), coagulation disorders, cardiovascular disease, respiratory disease, immune system disease, myocardial infarction, cardiac arrhythmia, obstructive or restrictive pulmonary disease.
3. Active tuberculosis (a history of tuberculosis exposure or a positive test for tuberculosis, including clinical, physical or imaging evidence).
4. Acute or chronic infectious diseases (including: syphilis or human T lymphoblast infection) (In this trial, patients with HIV, HTLV, or syphilis infection are also excluded. HIV-positive patients may have lower immunity, resulting in lower response to treatment or the toxicity after treatment is more sensitive)
5. Biliary or intestinal occlusion, cholangitis or severe gastrointestinal bleeding
6. Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease [SCID] and acquired immune deficiency syndrome [AIDS]).
7. ≥ grade 4 major organ immune-related Adverse Events (irAEs) following treatment with immune checkpoint inhibitors.
8. History of coronary revascularization or ischemic symptoms
9. Documented left ventricular ejection fraction (LVEF) of less than or equal to 45% tested in patients with:

   1. Clinically significant atrial and/or ventricular arrhythmias including but not limited to: atrial fibrillation, ventricular tachycardia, second or third degree heart block
   2. Age ≥ 60 years old
10. A rapidly deteriorating disease that the trial investigators believe not be able to tolerate treatment or testing procedures

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2021-04-09 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Acute, subacute toxicities and AEs of neoantigen-expanded autologous immune cell therapy. | Baseline to 20 weeks after cell infusion
  Number of participants with ≥ grade 3 immune related Adverse Events (irAEs) as assessed by CTCAE v6.0.
Dose-limiting toxicity (DLT) | Day 28
  Determination of DLT to be made after receiving the second dose of cell product of each cohort.
Maximum tolerated dose (MTD) | until Day 28
  The dose where no DLT is observed among 3 consecutive participants, or no more than one DLT among 6 participants.

SECONDARY OUTCOMES:
The antitumor activity of neoantigen-expanded autologous immune cell therapy | every 6 weeks up to 24 weeks after cell infusion.
  Number of participants with complete response and partial response, as s assessed by RECIST 1.1 and RANO.

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Mo Hou, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Linkou, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zacharakis N, Chinnasamy H, Black M, Xu H, Lu YC, Zheng Z, Pasetto A, Langhan M, Shelton T, Prickett T, Gartner J, Jia L, Trebska-McGowan K, Somerville RP, Robbins PF, Rosenberg SA, Goff SL, Feldman SA. Immune recognition of somatic mutations leading to complete durable regression in metastatic breast cancer. Nat Med. 2018 Jun;24(6):724-730. doi: 10.1038/s41591-018-0040-8. Epub 2018 Jun 4. PMID 29867227
- [Background] Chen F, Zou Z, Du J, Su S, Shao J, Meng F, Yang J, Xu Q, Ding N, Yang Y, Liu Q, Wang Q, Sun Z, Zhou S, Du S, Wei J, Liu B. Neoantigen identification strategies enable personalized immunotherapy in refractory solid tumors. J Clin Invest. 2019 Mar 5;129(5):2056-2070. doi: 10.1172/JCI99538. Print 2019 May 1. PMID 30835255
- See also: The protocol of this study is referenced by Zacharakis N et al. study. — https://pubmed.ncbi.nlm.nih.gov/29867227/
- See also: The protocol of this study is referenced by Chen F et al. study. — https://pubmed.ncbi.nlm.nih.gov/30835255/